CLINICAL TRIAL: NCT03655795
Title: Autologous Transplantation of Bronchial Basal Cells for Treatment of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Autologous Transplantation of Bronchial Basal Cells for Treatment of COPD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Regend Therapeutics (Industry)
Responsible Party: Principal Investigator, Jieming QU, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201809
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchial basal cells (Experimental): Autologous transplantation of bronchial basal cells
  Interventions: Biological: Bronchial basal cells

INTERVENTIONS:
Biological: Bronchial basal cells — Autologous transplantation of bronchial basal cells

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a disease characterized by long-term poor airflow, resulting in chronic pulmonary heart disease, chronic respiratory failure or even death. Till now, the damaged pulmonary bronchus structures in COPD patients cannot be repaired by recent clinical methods so far. In this study, we intends to carry out a single-centered, non-randomized and self-controlled clinical trial at an early phase. During the process, autologous bronchial basal cells (BBCs) will be dissected from trial tissue from bronchoscopic brushing. Then the BBCs will be expanded and detected by quality control. In the following, qualified BBCs will be injected directly into the lesion by fiberoptic bronchoscopy after lavage. After six-month observation, the investigators will evaluate the safety and effectiveness of the treatment by measuring a serial of indicators, including occurrence of adverse events, pulmonary function, the CT imaging, 6 minute walk distance (6MWD), St. George's Respiratory Questionnaire (SGRQ), modified medical research council (mMRC) dyspnea scale and COPD assessment test (CAT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 40 to 75.
* Subjects diagnosed with COPD and meet the following standards: a.sustained airway obstruction; b.presence of persistent airflow limitation confirmed by post-bronchodilator FEV1<70% predicted value and FEV1/FVC < 0.7.
* Subjects with pulmonary emphysema confirmed by imaging evidence.
* Subjects with DLCO<80% predicted value in pulmonary function test.
* Subjects with stable condition for more than 4 weeks.
* Subjects tolerant to bronchoscopy.
* Subjects signed informed consent.

Exclusion Criteria:

* Pregnant or lactating women.
* Subjects with syphilis or any of HIV, HBV, HCV positive antibody.
* Subjects with any malignancy.
* Subjects suffering from any of the following pulmonary diseases: asthma, active tuberculosis, pulmonary embolism, pneumothorax, pulmonary artery hypertension or interstitial lung disease.
* Subjects suffering from other serious diseases, such as diabetes, myocardial infarction, unstable angina, cirrhosis, and acute glomerulonephritis.
* Subjects with leukopenia (WBC less than 4x10^9 / L) or agranulocytosis (WBC less than 1.5x10^9 / L or neutrophils less than 0.5x10^9 / L) caused by any reason.
* Subjects with severe renal impairment, serum creatinine> 1.5 times of the upper limit of normal.
* Subjects with liver disease or liver damage: ALT, AST, total bilirubin> 2 times of the upper limit of normal.
* Subjects with a history of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders.
* Subjects with severe arrhythmias (such as ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter, etc.) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG.
* Subjects with a history of alcohol or illicit drug abuse.
* Subjects accepted by any other clinical trials within 3 months before the enrollment.
* Subjects with poor compliance, difficult to complete the study.
* Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Diffusing capacity of the lung for carbon monoxide (DLCO) | 6 months -1 year
  An indicator for pulmonary function

SECONDARY OUTCOMES:
Forced expiratory volume measured at the first second (FEV1) | 6 months -1 year
  One of the indicators in pulmonary function test, a marker to assess airway obstruction
Forced vital capacity (FVC) | 6 months -1 year
  One of the indicators in pulmonary function test, indicating the maximum amount of air a person can expel from the lungs after a maximum inhalation
The ratio of forced expiratory volume in the first one second to the forced vital capacity (FEV1/FVC) | 6 months -1 year
  One of the indicators in pulmonary function test, representing the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration to the full vital capacity
Maximum Mid Expiratory Flow (MMF) | 6 months -1 year
  One of the indicators in pulmonary function test, standing for maximal (mid-)expiratory flow and is the peak of expiratory flow as taken from the flow-volume curve and measured in liters per second
Maximum Voluntary Ventilation (MVV) | 6 months -1 year
  One of the indicators in pulmonary function test, measuring the maximum amount of air that can be inhaled and exhaled within one minute
6-minute-walk test (6MWT) | 6 months -1 year
  An indicator to evaluate the exercise function of patients with moderate or severe pulmonary heart diseases
Imaging of lung structure by high resolution computed tomography (HR-CT) | 6 months -1 year
  Images of lung will be analyzed to indicate the newly-derived pulmonary structure.
Assess life quality affected by the respiratory problem by St. George's respiratory questionnaire (SGRQ) scale | 6 months -1 year
  Total scores (0-100) will be calculated and compared before and after transplantation, and higher values represent a better outcome.
Modified medical research council (mMRC) chronic dyspnea scale to evaluate the level of dyspnea | 6 months -1 year
  mMRC Dyspnea Scale scores (1-5) will be measured and compared before and after transplantation, and lower values represent a better outcome.
COPD Assessment Test (CAT) | 6 months -1 year
  A patient-completed questionnaire assessing all aspects of the impact of COPD

CONTACTS AND LOCATIONS:
Overall Officials: Yun Feng, M.D., Ph.D, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuo W, Zhang T, Wu DZ, Guan SP, Liew AA, Yamamoto Y, Wang X, Lim SJ, Vincent M, Lessard M, Crum CP, Xian W, McKeon F. p63(+)Krt5(+) distal airway stem cells are essential for lung regeneration. Nature. 2015 Jan 29;517(7536):616-20. doi: 10.1038/nature13903. Epub 2014 Nov 12. PMID 25383540
- [Background] Ma Q, Ma Y, Dai X, Ren T, Fu Y, Liu W, Han Y, Wu Y, Cheng Y, Zhang T, Zuo W. Regeneration of functional alveoli by adult human SOX9+ airway basal cell transplantation. Protein Cell. 2018 Mar;9(3):267-282. doi: 10.1007/s13238-018-0506-y. Epub 2018 Jan 17. PMID 29344809